CLINICAL TRIAL: NCT05976802
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose Ranging Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Budesonide Rectal Foam BID for 2 Weeks, Followed by QD for 4 Weeks, in Pediatric Patients Aged 5 to 17 Years With Active, Mild to Moderate Distal Ulcerative Colitis
Brief Title: Dose Ranging Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Budesonide Rectal Foam in Pediatric Patients Aged 5 to 17 Years With Active, Mild to Moderate Distal Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFUC4991
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose budesonide rectal foam (Experimental)
  Interventions: Drug: High dose budesonide rectal foam
- Low dose budesonide rectal foam (Experimental)
  Interventions: Drug: Low dose budesonide rectal foam
- Matching placebo rectal foam (Placebo Comparator)
  Interventions: Drug: Matching placebo rectal foam

INTERVENTIONS:
Drug: High dose budesonide rectal foam — Twice a day for 2 weeks, then once a day for 4 weeks
  Arms: High dose budesonide rectal foam
Drug: Low dose budesonide rectal foam — Twice a day for 2 weeks, then once a day for 4 weeks
  Arms: Low dose budesonide rectal foam
Drug: Matching placebo rectal foam — Twice a day for 2 weeks, then once a day for 4 weeks
  Arms: Matching placebo rectal foam

SUMMARY:
The primary objective of this study is to evaluate the efficacy (as measured by induction of remission) of two dose levels (low and high) per age group (5 to <12 and 12 to ≤17 years) of budesonide rectal foam as compared to an equivalent volume of rectally administered placebo foam over the same dosing schedule, in pediatric subjects with active, mild to moderate distal ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female (non-pregnant and non-lactating) 5 to ≤17 years of age at Screening.
2. Established diagnosis of UC, based on clinical history, characteristic endoscopic findings, and histopathology results from biopsies.
3. Disease limited to the distal colon and rectum, (disease involving only the first 15 centimeters or less proximal to the anal verge).
4. Active, distal UC of mild or moderate severity, defined as a Modified Mayo Clinic Score (mMCS) between 4 and 8, inclusive, that includes an endoscopy subscore ≥ 2 and a rectal bleeding subscore ≥ 1.
5. If on a background oral 5-ASA, the dose and formulation have remained unchanged for at least 6 weeks prior to Visit 2 (Run-In) and the subject is willing to remain on the same dosage form and regimen for the duration of the study.

Exclusion Criteria:

1. Current or prior diagnosis of Crohn's disease or indeterminate colitis.
2. Ulcerative colitis involving the proximal colon - i.e, the sigmoid, left, transverse, and/or ascending colon and cecum;
3. Severe UC, defined as an mMCS > 8.
4. Infectious colitis (based on positive microbiologic tests at Screening) or any recent history of infectious colitis (within 30 days of Screening).
5. Prior gastrointestinal surgery, except appendectomy or hernia (e.g., inguinal, umbilical).

   NOTE: Prior cholecystectomy is not exclusionary if more than 1 year prior to Screening.
6. Evidence or history of toxic megacolon or bowel resection.
7. Active proctologic pathology such as hemorrhoids, fistulas and fissures or other historical anatomic problems which would impair rectal administration (e.g., cloaca, imperforate anus history)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2027-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with clinical remission | Day 42
  Clinical remission based on the modified Mayo Clinic Score, defined as an endoscopy score ≤ 1 (excluding friability), a rectal bleeding subscore of 0, and at least a 1-point decrease in stool frequency subscore from Baseline to achieve a stool frequency subscore ≤ 1. Each component is scored from 0 to 3, with total scores ranging from 0 to 9, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Proportion of participants who achieve a rectal bleeding subscale score of 0 at the end of six weeks of treatment | Day 42
  Scored from 0 to 3, with higher scores indicating more severe disease.
Proportion of participants who achieve a stool frequency subscale score of 0 at the end of six weeks of treatment. | Day 42
  Scored from 0 to 3, with higher scores indicating more severe disease.
Proportion of subjects who achieve an endoscopy subscale score of 0 or 1 at the end of six weeks of treatment. | Day 42
  Scored from 0 to 3, with higher scores indicating more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health

IPD SHARING:
Plan to Share IPD: Undecided